CLINICAL TRIAL: NCT04444739
Title: AtrophyLSS - Association Between Lumbar Muscle Atrophy, Sagittal Pelvic Alignment and Stenosis Grade in Patients With Degenerative Lumbar Spinal Stenosis
Brief Title: Association Between Lumbar Muscle Atrophy, Sagittal Pelvic Alignment and Stenosis Grade in Patients With Degenerative Lumbar Spinal Stenosis
Acronym: AtrophyLSS
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00150; ch20Muendermann4
Record Dates: First submitted 2020-06-16; First posted 2020-06-24 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Lumbar Spinal Stenosis (LSS)
Keywords: paraspinal muscle atrophy (MA); sagittal pelvic alignment; degenerative spine diseases; stenosis grade (SG); degenerative LSS; Goutallier classification
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: radiographic data collection — From existing radiological Images (upright standing X-ray and supine MRI of the lumbar spine), specific radiographic parameters will be extracted

SUMMARY:
This study is to evaluate the correlation between muscle atrophy (MA), sagittal alignment, and stenosis degree in patients with lumbar spinal Stenosis (LSS). From existing radiological images, specific radiographic parameters will be extracted. General Information (Age, sex, levels of stenosis, duration of symptoms) will be extracted from patient files.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of degenerative lumbar spinal stenosis
* Upright standing sagittal plane X-ray of lumbar spine with clear visibility of pelvis sacrum and femoral head
* MRI of the lumbar region with clear visibility of different muscle atrophy grade
* Consent that health related information can be used for research was signed

Exclusion Criteria:

* Other spinal disease such as severe scoliosis, fracture, spondylolisthesis and ankylosing spondylitis.
* Neuromuscular diseases such as M.Parkinson or multiple sclerosis
* Previous surgery of the spine
* Infection and/or malignancy tumor with involvement of the bony or soft tissue structures of the spine
* Presence of a documented consent dissent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who visited Orthopaedics and Traumatology outpatient clinic at University Hospital Basel for clinical and radiological consultation regarding their lumbar spine between 01.01.2018 and 31.12.2019.
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Severity of muscle atrophy (MA) from supine Magnetic Resonance Imaging (MRI) of lumbar spine | single time-point at baseline
  Muscle atrophy stage will be observed using Goutallier classification
  * Stage 0: No fatty infiltration
  * Stage 1: Few fatty streaks within the muscle
  * Stage 2: Less than 50% fat within the muscle
  * Stage 3: 50% of fat within the muscle
  * Stage 4: more than 50% fat with in the muscle. The MA stage will be observed in MRI of 5 lumbar disc levels (L1-S1). The MA stage of patients will be calculated as average stage of five lumbar segments.
Pelvic incidence (PI): Pelvic alignment from standard upright standing sagittal plane X-ray of lumbar spine with clear visibility of pelvis sacrum and femoral heads | single time-point at baseline
  Pelvic incidence (PI): The angle between the line perpendicular to the sacral endplate at its midpoint and a line connecting this point to the axis of the femoral head.
Severity of stenosis from supine MRI of lumbar spine | single time-point at baseline
  Stenosis grade will be observed using Schizas classification (Schizas et al., 2010)
  * Grade 1: Dural sac party occupied by the rootlets; Cerebrospinal fluid clearly visible; No stenosis
  * Grade 2: Rootlets occupy whole dural sac; Some cerebrospinal fluid visible; Moderate stenosis.
  * Grade 3: Rootlets not visible; No cerebrospinal fluid visible; Epidural fat posteriorly; Severe stenosis.
  * Grade 4: Rootlets not visible; No cerebrospinal fluid; No epidural fat; Extreme Stenosis. The most severe level will be regarded as the stenosis grade of the patients.
Pelvic tilt (PT): Pelvic alignment from standard upright standing sagittal plane X-ray of lumbar spine with clear visibility of pelvis sacrum and femoral heads | single time-point at baseline
  Pelvic tilt (PT): The angle formed by a vertical line through the center of the femoral heads and the line from the center of the femoral axis and the midpoint of the sacral end plate.
Sacral slope (SS): Pelvic alignment from standard upright standing sagittal plane X-ray of lumbar spine with clear visibility of pelvis sacrum and femoral heads | single time-point at baseline
  Sacral slope (SS): The angle formed between the horizontal and the sacral end plate.
Lumbar lordosis (LL): Pelvic alignment from standard upright standing sagittal plane X-ray of lumbar spine with clear visibility of pelvis sacrum and femoral heads | single time-point at baseline
  Lumbar lordosis (LL): The sagittal angle formed between the superior end plate of L1 and the sacral end plate

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Muendermann, Prof. Dr. med., Principal Investigator — Orthopaedics and Traumatology, University Hospital Basel
Locations (1):
- Orthopaedics and Traumatology, University Hospital Basel, Basel, Switzerland